CLINICAL TRIAL: NCT04312035
Title: Effect of End-range Mobilization in Addition to Conservative Therapy on Decrease of Pressure Pain Threshold
Brief Title: Effect of Combined Interventions on Pressure Pain Threshold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML_PPT_PhysTher
Record Dates: First submitted 2020-03-04; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Osteo Arthritis Knee
Keywords: Musculoskeletal Manipulations; Osteoarthritis, Knee; Pain Threshold; Conservative Treatment
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- End-range mobilization (Experimental): End-range mobilization performed in end-position of the knee joint
  Interventions: Procedure: end-range mobilization
- Non end-range mobilization (Experimental): Non end-range mobilization performed in loose-packed position of the knee joint
  Interventions: Procedure: Non end-range mobilization
- Control (Placebo Comparator): Sham technique performed in loose-packed position of the knee joint
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: end-range mobilization — accessory technique applied on the tibiofemoral joint with the aim of increasing extensibility of the periarticular tissues
  Arms: End-range mobilization
Procedure: Non end-range mobilization — accessory technique applied on the tibiofemoral joint with the aim of alleviating pain
  Arms: Non end-range mobilization
Procedure: Control — hands-on cutaneous technique
  Arms: Control

SUMMARY:
The effect of mobilizations on decrease of peripheral and central sensitivity has been proven in KOA. Furthermore, the effect of conservative therapy has also been proven in the increase of pain threshold in KOA. However, no study has investigated the effect of these interventions combined till date in KOA.

The aim of the present study is to investigate the short-term and long-term effect of end-range mobilization in addition to conservative therapy on decrease of pressure pain threshold in KOA.

DETAILED DESCRIPTION:
The positive effect of different manual mobilizations have been proven in the management of knee osteoarthritis (KOA). Pressure pain threshold, as a measure of somatosensory function, is a well-applied measurement technique for the pain perception in KOA. The effect of mobilizations on decrease of peripheral and central sensitivity has been proven in KOA. Furthermore, few studies has revealed the effect of conservative therapy as an effective intervention in the increase of pain threshold. However, no study has investigated the effect of these interventions combined till date in KOA, which could give a long-lasting effect in the decrease of sensitization in KOA.

Therefore, the aim of the present study is to investigate the short-term and long-term effect of end-range mobilization in addition to conservative therapy on decrease of pressure pain threshold in KOA.

ELIGIBILITY:
Inclusion Criteria:

* clinical classification criteria of knee osteoarthritis according to the American College of Rheumatology
* categorization as End of Range Problem based on Maitland manual therapy
* unilateral/bilateral moderate-to-severe symptomatic tibiofemoral KOA with radiographic evidence of Kellgren-Lawrence scale 2 or 3
* pain during weight-bearing activities at least within 6 months
* at least 90° knee flexion
* sufficient mental status

Exclusion Criteria:

* acute inflammation of the knee
* total knee replacement in the opposite side
* class II. obesity (body mass index>35kg/m2)
* severe degenerative lumbar spine disease (e.g. spondylolisthesis)
* systemic inflammatory arthritic or neurological condition
* physiotherapy/balneotherapy attendance or manual therapy within 3 months
* intraarticular injections in the prior 12 months
* use of walking aid
* contraindication for manual therapy
* complex regional pain syndrome
* cognitive impairment

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
change of peripheral sensitivity | following 3-week rehabilitation
  peripheral sensitivity (pressure pain threshold) assessed at the local knee
change of peripheral sensitivity | following 3-month
  peripheral sensitivity (pressure pain threshold) assessed at the local knee

SECONDARY OUTCOMES:
change of central sensitivity | following 3-week rehabilitation
  central sensitivity (pressure pain threshold) assessed at the ipsilateral m. extensor carpi radialis longus
change of central sensitivity | following 3-month
  central sensitivity (pressure pain threshold) assessed at the ipsilateral m. extensor carpi radialis longus
change of general pain intensity | following 3-week rehabilitation
  general pain intensity from the previous week using the Visual Analogue Scale
change of general pain intensity | following 3-month
  general pain intensity from the previous week using the Visual Analogue Scale
change of Timed Up and Go test | following 3-week rehabilitation
  short test for measuring physical performance
change of Timed Up and Go test | following 3-month
  short test for measuring physical performance
change of pain intensity during physical performance | following 3-week rehabilitation
  pain intensity measured during the previously mentioned physical performance test using the 0-10 Numerating Pain Rating Scale, where 0 indicate no pain and 10 indicate worst imaginable pain
change of pain during physical performance | following 3-month
  pain intensity measured during the previously mentioned physical performance test using the 0-10 Numerating Pain Rating Scale, where 0 indicate no pain and 10 indicate worst imaginable pain
degree of knee flexion during passive movement at the onset of knee pain | following 3-week rehabilitation
  measurement of degree of knee flexion during passive movement at the onset of knee pain
degree of knee flexion during passive movement at the onset of knee pain | following 3-month
  measurement of degree of knee flexion during passive movement at the onset of knee pain
strength of resistance of passive knee flexion at the onset of knee pain | following 3-week rehabilitation
  measurement of strength of resistance arising from the anterior located tissues around the knee during passive knee flexion at the onset of pain
strength of resistance of passive knee flexion at the onset of knee pain | following 3-month
  measurement of strength of resistance arising from the anterior located tissues around the knee during passive knee flexion at the onset of pain

CONTACTS AND LOCATIONS:
Overall Officials: Miklós Pozsgai, MSc, Principal Investigator — Zsigmondy Vilmos Spa and Balneological Hospital of Harkány
Locations (1):
- Miklós Pozsgai, Harkány, Please Select, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McAlindon TE, Bannuru RR, Sullivan MC, Arden NK, Berenbaum F, Bierma-Zeinstra SM, Hawker GA, Henrotin Y, Hunter DJ, Kawaguchi H, Kwoh K, Lohmander S, Rannou F, Roos EM, Underwood M. OARSI guidelines for the non-surgical management of knee osteoarthritis. Osteoarthritis Cartilage. 2014 Mar;22(3):363-88. doi: 10.1016/j.joca.2014.01.003. Epub 2014 Jan 24. PMID 24462672
- [Background] Bajaj P, Bajaj P, Graven-Nielsen T, Arendt-Nielsen L. Osteoarthritis and its association with muscle hyperalgesia: an experimental controlled study. Pain. 2001 Aug;93(2):107-114. doi: 10.1016/S0304-3959(01)00300-1. PMID 11427321
- [Background] Imamura M, Imamura ST, Kaziyama HH, Targino RA, Hsing WT, de Souza LP, Cutait MM, Fregni F, Camanho GL. Impact of nervous system hyperalgesia on pain, disability, and quality of life in patients with knee osteoarthritis: a controlled analysis. Arthritis Rheum. 2008 Oct 15;59(10):1424-31. doi: 10.1002/art.24120. PMID 18821657
- [Background] Moss P, Sluka K, Wright A. The initial effects of knee joint mobilization on osteoarthritic hyperalgesia. Man Ther. 2007 May;12(2):109-18. doi: 10.1016/j.math.2006.02.009. Epub 2006 Jun 13. PMID 16777467